CLINICAL TRIAL: NCT06280573
Title: COld Exposure With Controlled BReathing And Meditation in Patients With Multiple Sclerosis (COBRAMS)
Acronym: COBRAMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS1
Record Dates: First submitted 2024-01-23; First posted 2024-02-28 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Combination Product: Wim Hoff method
- control group (No Intervention)

INTERVENTIONS:
Combination Product: Wim Hoff method — breathing exercises, cold exposure, and meditation
  Arms: intervention group

SUMMARY:
The goal of this interventional study is to test the effect of the anti-inflammatory and neuroprotective effects of this supplementary training program that includes breathing exercises, cold exposure, and meditation in patients diagnosed with multiple sclerosis.

Researchers will compare the effect to control groups of MS patients without intervention.

ELIGIBILITY:
Inclusion Criteria:

* RRMS diagnosed according to the official 2020 McDonald's criteria,
* age 18-55 years,
* MS duration up to 10 years,
* EDSS 1.0-5.5,
* willingness to participate

Exclusion Criteria:

* relapse or corticosteroid treatment within 3 months prior to study enrollment
* severe/unstable comorbidity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
concentration of pro-inflammatory cytokines | 12 weeks
  blood concentrations in pg/ml of
  • cytokines (interleukins - IL-1β, IL-6, IL-8, IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33, interferons IFN-α2 and IFN-γ, tumor necrosis factor TNF-α, monocyte chemoattractant protein MCP-1)
concentration of markers of oxidative stress | 12 weeks
  blood concentration in mmol/l of markers of oxidative stress (OS) - advanced glycation end products (AGEs), fructosamine, advanced oxidation protein products (AOPP), thiobarbituric acid reactive substances (TBARS), total antioxidant capacity (TAC), ferric reducing ability of plasma (FRAP),
concentration of NfL | 12 weeks
  neurofilamen light chains
concentration of GFAP | 12 weeks
  glial fibrillary acidic protein
concentration of ecDNA | 12 weeks
  cell-free extracellular DNA

SECONDARY OUTCOMES:
Expanded Disability Status Scale | 12 weeks
  physical disability - score from 0.0 to 10.0
Timed 25-Foot Walk | 12 weeks
  walking speed in seconds
Nine-Hole Peg Test | 12 weeks
  finger dexterity in seconds
Symbol Digit Modalities Test | 12 weeks
  cognitive status - score in 90s
Fatigue Scale for Motor and Cognitive Functions | 12 weeks
  to assess multiple sclerosis-related fatigue
General Anxiety Disorder-7 | 12 weeks
  level of anxiety
Patient Health Questionnaire-9 | 12 weeks
  assesses degree of depression severity

CONTACTS AND LOCATIONS:
Locations (1):
- Derer's University Hospital, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No